CLINICAL TRIAL: NCT00453271
Title: A Randomized, Double-Blind, Parallel-Group,Multicenter, Dose-Response, Vehicle-Controlled Study of the Safety and Efficacy of NB-002 in the Treatment of Mild to Moderate Distal Subungual Onychomycosis of the Toenail
Brief Title: Treatment of Mild to Moderate Distal Subungual Onychomycosis of the Toenail
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NanoBio Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NB-002-002
Record Dates: First submitted 2007-03-26; First posted 2007-03-28 (Estimated); Last update posted 2013-05-23 (Estimated); Status verified 2013-05

CONDITIONS: Onychomycosis
Keywords: chronic persistent infection of the nail bed or plate
MeSH Terms: conditions — Onychomycosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- NB-002 0.25% BID (Experimental)
  Interventions: Drug: NB-002
- NB-002 0.5% QD (Experimental)
  Interventions: Drug: NB-002
- NB-002 0.5% BID (Experimental)
  Interventions: Drug: NB-002
- Vehicle control (Sham Comparator)
  Interventions: Drug: Vehicle control

INTERVENTIONS:
Drug: NB-002
  Arms: NB-002 0.25% BID; NB-002 0.5% BID; NB-002 0.5% QD
Drug: Vehicle control
  Arms: Vehicle control

SUMMARY:
The purpose of the study is to determine whether NB002, 0.25%, and 0.5% are safe and effective in the treatment of distal subungual onychomycosis of the toenail.

DETAILED DESCRIPTION:
The purpose of the study is to determine whether NB002, 0.25%, and 0.5% are safe and effective in the treatment of distal subungual onychomycosis of the toenail.

ELIGIBILITY:
Inclusion Criteria:

* are healthy males or females between the ages of 18 and 75 years of age;
* have a clinical diagnosis of mild to moderate DSO in the nail of at least one great toe, involving 25%-67% of the nail, without lunular or proximal involvement;
* positive mycology results (ie, KOH test and culture of a dermatophyte) from the target great toenail;
* refrain from using any lotions, creams, liquids, or polish on treated toenails or on the skin immediately adjacent to the toenails during the treatment period unless directed to do so by the investigator;
* are willing to refrain from using topical steroids or topical antifungals on toenails or the skin immediately adjacent to the toenails; or systemic antifungals for the duration of the study;

Exclusion Criteria:

* females who are pregnant, plan to become pregnant during the study, or are nursing a child;
* are hypersensitive to topical creams, ointments, medications, or surfactants;
* have received systemic antifungal therapy for any reason within 3 months, or topical antifungal therapy on the toenails or skin immediately adjacent to the toenails within 3 weeks prior to the start of the study; or
* have taken any investigational drug within 4 weeks prior to the start of the study.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 443 (Actual)
Dates: Start 2007-01; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Planimetry assessment of the target great toenail | Week 24
Rate of complete cure | Week 46
Rate of therapeutic success | Week 46

SECONDARY OUTCOMES:
Investigator's visual assessment of length of new unaffected nail
The presence/absence of DSO on all toenails

CONTACTS AND LOCATIONS:
Overall Officials: Alicia Barba, MD, Principal Investigator — International Dermatology Research, Inc.; Alicia Bucko, DO, Principal Investigator — Academic Dermatology Associates; Richard Pollak, DPM, MS, Principal Investigator — Endeavor Clinical Trials, PA; Michael Jarratt, MD, Principal Investigator — Derm Research, PLLC; Terry Jones, MD, Principal Investigator — J & S Studies, Inc.; Robert Kaylor, DPM, Principal Investigator — Welborne Clinic; Steven Kempers, MD, Principal Investigator — Minnesota Clinical Study Center; Robert Matheson, MD, Principal Investigator — Oregon Medical Research Center, PC; Brock McConnehey,, DO, Principal Investigator — Northwest Clinical Trial; David Pariser, MD, Principal Investigator — Virginia Clinical Research, Inc.; Phoebe Rich, MD, Principal Investigator — Oregon Dermatology and Research Center; Dan Stewart, DO, Principal Investigator — Michigan Center for Research Corp; Leonard Swinyer, MD, Principal Investigator — Dermatology Research Center, Inc.; Robert Bissonette, MD, Principal Investigator — Innovaderm Research Inc.; Sylvia Garnis-Jones, MD, Principal Investigator — EntraLogix Clinical Group Inc.; David Gratton, MD, Principal Investigator — International Dermatology Research, Inc.; Lyn Guenther, MD, Principal Investigator — The Guenther Dermatology Research Centre; Rod Kunynetz, MD, Principal Investigator — Ultranova Skincare; Charles Lynde, MD, Principal Investigator — Lynderm Research, Inc.; Richard Langley, MD, Principal Investigator — Eastern Canada Cutaneous Research Associates, LTD; Kim Papp, MD, Principal Investigator — K. Papp Clinical Research; Yves Poulin, MD, Principal Investigator — Centre de Reeberche Dermatologique du Quebec Metropolitain (CRDQ); Wayne Gulliver, MD, Principal Investigator — Newlab Clinical Research Inc.; R G Sibbald, MD, Principal Investigator — Dermatology Clinic
Locations (24):
- United States (13):
  - International Dermatology Research, Miami, Florida
  - Northwest Clinical Trial, Boise, Idaho
  - Welborne Clinic, Evansville, Indiana
  - Michigan Center for Research Corp., Clinton Township, Michigan
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - Academic Dermatology Associates, Albuquerque, New Mexico
  - Oregon Dermatology and Research Center, Portland, Oregon
  - Oregon Medical Research Center, PC, Portland, Oregon
  - DermResearch Inc., Austin, Texas
  - J & S Studies, Inc., Bryan, Texas
  - Endeavor Clinical Trials, PA, San Antonio, Texas
  - Dermatology Research Center, Inc., Salt Lake City, Utah
  - Virginia Clinical Research, Inc., Norfolk, Virginia
- Canada (11):
  - Newlab Clinical Research, Inc., St. John's, Newfoundland and Labrador
  - Eastern Canada Cutaneous Research Associates, LTD, Halifax, Nova Scotia
  - Ultranova Skincare, Barrie, Ontario
  - The Guenther Dermatology Research Centre, London, Ontario
  - Lynderm Research, Inc., Markham, Ontario
  - Dermatology Clinic, Mississauga, Ontario
  - EntraLogix Clinical Group, Inc., Oakville, Ontario
  - K. Papp Clinical Research, Waterloo, Ontario
  - Innovaderm Research, Inc., Montreal, Quebec
  - International Dermatology Research, Inc., Montreal, Quebec
  - Centre de Reeberche Dermatologique du Quebec Metropolitain (CRDQ), Québec, Quebec